CLINICAL TRIAL: NCT00872313
Title: Potential Risk Factors for Postpartum Psychosis
Brief Title: Risk Factors for Postpartum Psychosis
Acronym: RIFPP
Status: Completed | Type: Observational
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Fu Zhou Wang, Dr, Nanjing Medical University
Other Study IDs: NMU-200903-MZ003; NJFY09102M107
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Postpartum Period; Psychosis
Keywords: Labor; Psychology; Postpartum Psychology
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Psychoses within the first 3 months postpartum
- 2: Psychoses > 3 months to 6 months postpartum

SUMMARY:
A range of psychological disorders occur in women in the postpartum period. These include "the blues", which occurs in the first days after birth and which is very common and self-limiting; severe psychoses often associated with mania or bipolar illness, occurring in the first weeks after birth; and mild to moderate depression, occurring weeks to months after birth. Studies have been done focused on postpartum psychosis using a retrospective investigation, which gave only a limited material on the prevalence of psychological disorders in postpartum women. The investigators hypothesized that different pathways to psychosis function as the risk factors which may be overlapped, truly independent, mediating, or moderating, in new mothers who are at high risk and/or during the early period of delivery. In addition, the investigators purposed that the temporal sequence of biological, social and demographic variables are also the potential factors contributing to the development of postpartum psychosis.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Chinese

Exclusion Criteria:

* Age < 18 years or > 50 years
* Gestational age < 32 weeks

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Parturients undergoing spontaneous or induced labor or cesarean delivery
Sampling Method: Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2009-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Incidence of psychoses | 3 months and 6 months postpartum

SECONDARY OUTCOMES:
Antepartum economic level | One year before labor and delivery (recorded by antepartum communication)
Antepartum social status | One year before labor and delivery (recorded by antepartum communication)
Antepartum psychological level | 1 day before birth
Intrapartum complications | 1 day after birth
Baby characteristics | One minute, 5min, 15min after baby was born
Maternal characteristics | One day after birth
Medical caregiver characteristics | One day before and after the labor completion
Parturient family characteristics | One week before labor and delivery, recorded by investigators through patients' antepartum communication
Intrapartum medical procedures | One day after birth

CONTACTS AND LOCATIONS:
Overall Officials: XiaoFeng Shen, MD, Study Director — Nanjing Medical University
Locations (1):
- Nanjing Maternal and Child Health Care Hospital, Nanjing, Jiangsu, China